CLINICAL TRIAL: NCT00074789
Title: Reducing Depressive Symptoms in Low-Income Mothers
Brief Title: Reducing Symptoms of Depression in Low-Income Mothers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linda Beeber, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH065524 (NIH); R01MH065524 (NIH); DSIR 83-ATAS; HILDA
Record Dates: First submitted 2003-12-19; First posted 2003-12-22 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Early Head Start Program
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive home-based interpersonal depression treatment for 26 weeks
  Interventions: Behavioral: Modified Interpersonal Therapy
- 2 (Active Comparator): Participants will receive attention control/usual care for 26 weeks
  Interventions: Behavioral: Attention control/usual care

INTERVENTIONS:
Behavioral: Modified Interpersonal Therapy — Psychiatric mental health nurses will meet with participants 10 times, an hour each time, over a period of 14 weeks. The nurses will continue to work with the mothers over the next 8 weeks by phone, conducting 5 fifteen minute phone sessions.
  Arms: 1
Behavioral: Attention control/usual care — Participants will receive the usual care for depression.
  Arms: 2

SUMMARY:
This study will test the effectiveness of a short-term intervention in treating depressed young mothers with young children enrolled in Early Head Start Programs.

DETAILED DESCRIPTION:
Limited resources, poor social support, and complex life problems contribute to the high prevalence and severity of depressive symptoms in low-income mothers. As depressive symptoms persist, they often rob young mothers of the energy they need for school, job training, and positive interaction with their children, which can negatively affect a child's language acquisition, intellectual development, and social conduct. This study will design and implement a home-based treatment to help young mothers manage their depressive symptoms, increase their social support, manage or resolve life issues, and effectively parent their infant or toddler through the use of EHS resources.

Mothers will be randomly assigned to receive either home-based interpersonal depression treatment or an attention control/usual care condition for 26 weeks. Assessments will be made at study start and Weeks 14, 22, and 26. Depression scales, interviews, and analyses of videotaped mother-child interactions will be used to assess participants. Stress, social support, and use of EHS services will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Score of 16 or higher on the Center for Epidemiological Studies Depression (CES-D) Scale
* Child who is 6 weeks to 30 months old
* Child who is enrolled in an Early Head Start program

Exclusion Criteria:

* Regular use of psychotropic medication
* Regular use of psychotherapy or drug/alcohol treatment

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2003-06; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Level of depressive symptoms | Measured at Week 26

SECONDARY OUTCOMES:
Mother child interactions | Measured at Week 26

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - P.E.A.C.E, Inc. Early Head Start, Syracuse, New York
  - Asheville City Schools Preschool-Early Head Start Program, Asheville, North Carolina
  - Chapel Hill Training Outreach Project, Inc. Early Head Start, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - W.A.G.E.S., Inc. Early Head Start Program, Goldsboro, North Carolina
  - United Child Development Services, Inc. Early Head Start, Greensboro, North Carolina

REFERENCES:
- [Derived] Salomon RE, Muscatell KA, Crandell J, Anderson RA, Beeber LS. A Preliminary Investigation of Psychoneurological Symptoms in Low-Income Mothers. Nurs Res. 2021 Set/Oct 01;70(5):325-333. doi: 10.1097/NNR.0000000000000518. PMID 33935214